CLINICAL TRIAL: NCT04095208
Title: Combination of Nivolumab Plus Relatlimab in Patients With Advanced or Metastatic Soft-tissue Sarcoma: a Proof-of-concept Randomized Phase II Study.
Acronym: CONGRATS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2019-03; 2019-002332-81 (EudraCT Number); CA224-085 (Other: BMS)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Soft Tissue Sarcoma Adult; Advanced Cancer
Keywords: soft-tissue sarcoma; tertiary lymphoid structure; immunotherapy; oncology; metastatic
MeSH Terms: conditions — Sarcoma; Tertiary Lymphoid Structures; Neoplasms; Neoplasm Metastasis | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Randomized phase II trial - Arm A (Experimental): Combination of nivolumab and relatlimab.
  Interventions: Drug: Association of Nivolumab + Relatlimab
- Experimental: Randomized phase II trial - Arm B (Experimental): Treatment by nivolumab alone.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Association of Nivolumab + Relatlimab — A treatment cycle consists of 4 weeks.
  Nivolumab will be administered as a 30-minutes intravenous infusion, on Days 1 and 15 of each cycle (every 2 weeks) - [240 mg].
  Relatlimab will be administered as a 60-minutes intravenous infusion, on Days 1 and 15 of each cycle (every 2 weeks) - [80 mg].
  Arms: Experimental: Randomized phase II trial - Arm A
Drug: Nivolumab — A treatment cycle consists of 4 weeks.
  Nivolumab will be administered as a 30-minutes intravenous infusion, on Days 1 and 15 of each cycle (every 2 weeks) - [240 mg].
  Arms: Experimental: Randomized phase II trial - Arm B

SUMMARY:
This is a multicenter study assessing the efficacy of nivolumab in association with relatlimab.

DETAILED DESCRIPTION:
This multicenter, prospective, open-labeled 2-arm, randomized non-comparative phase II trial. This phase II trial is based on a 2-stage Simon's optimal design. Randomization 1:1 with 1 patient randomized in experimental arm A (association of nivolumab plus relatlimab) and 1 patient randomized in arm B (treatment by nivolumab alone).

ELIGIBILITY:
Inclusion Criteria:

1. Histology: participant with soft tissue sarcoma histologically confirmed and reviewed by the RRePS Network as recommended by the French NCI (Inca),
2. Presence of mature tertiary lymphoid structures (TLS). Except if presence of TLS have been already confirmed by Biopathological platform at Bergonié Institute, presence of TLS should be confirmed by central review based on FFPE (Formalin-Fixed Paraffin-Embedded) tumor tissue sample (archived or newly obtained by biopsy for research purpose). Note that the presence of TLS could be determined by central analysis if not available before,
3. Deleted MSA5
4. For research purpose, have provided tissue of a tumor lesion from < 3 months old archival tissue sample (both frozen or FFPE) obtained on locally advanced disease, or metastasis, with no subsequent treatment since or presence of tumor lesion that can be biopsied,
5. Advanced non resectable / metastatic disease,
6. Documented progression according to RECIST criteria, unless the participant has no received prior systemic treatment for advanced disease. Progression on the last line of treatment should be confirmed by central review with two radiological assessments identical (CT scans or MRI) obtained at less than 6 months interval within the 12 months before inclusion.
7. At least one tumor site that can be biopsied for research purpose,
8. Previous treatment: no more than 2 previous lines of systemic therapy for advanced or metastatic disease
9. Participant must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement,
10. Age ≥ 18 years,
11. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1,
12. Measurable disease according to RECIST v1.1 outside any previously irradiated field (except if progressive as per RECIST v1.1 at inclusion). At least one site of disease must be uni-dimensionally ≥ 10 mm,
13. Life expectancy > 3 months,
14. No symptomatic central nervous system disease,
15. No chronic use of glucocorticoids higher than 10 mg/day prednisone equivalent,
16. Adequate hematological, renal, metabolic and hepatic function:

    1. Hemoglobin > 9 g/dl (patients may have received prior red blood cell [RBC] transfusion, if clinically indicated); leucocytes ≥ 2 G/l, absolute neutrophil count (ANC) > 1.5 G/l and platelet count > 100 G/l, lymphocyte count > 0.5 G/l
    2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normality (ULN) (< 5 in case of liver metastasis).
    3. Total bilirubin < 1.5 x ULN OR Direct bilirubin < ULN for subjects with total bilirubin levels > 1.5 x ULN.
    4. Albumin > 25g/l.
    5. Serum creatinine < 1.5 x ULN OR Calculated creatinine clearance (CrCl) > 60 ml/min (calculated per institutional standard) for subject with creatinine levels > 1.5 x ULN.
    6. INR < 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    7. aPTT ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants,
    8. Thyroid functions (T3, T4 and TSH) ≤ 1.5 x ULN and ≥ LLN,
17. Left ventricular ejection fraction (LVEF) ≥ 50% assessed by TTE or MUGA (TTE preferred test) within 6 months from study entry,
18. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
19. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy, except for TKI which should be discontinued for > 2 weeks before treatment start
20. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2 (according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE, version 5.0),
21. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to study entry. Pregnancy test should be repeated within 24 hours prior to receiving the first dose of study medication.
22. Women must agree to use a medically acceptable method of contraception throughout the treatment period and for 6 months after discontinuation of treatment. Men must agree to use a medically acceptable method of contraception throughout the treatment period and for 8 months after discontinuation of treatment. Acceptable methods for contraception include intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year.
23. Voluntary signed and dated written informed consents prior to any specific study procedure,
24. Patients with a social security in compliance with the French law

Exclusion Criteria:

1. Previous treatment with an PD1/PDL1, LAG-3
2. Previous enrolment in the present study,
3. Evidence of progressive or symptomatic central nervous system (CNS) or leptomeningeal metastases,
4. Women who are pregnant or breast feeding,
5. Participant unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
6. Known hypersensitivity to any involved study drug or of its formulation components,
7. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
8. Uncontrolled cardiac arrhythmia or hypertension, as per investigator discretion,
9. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

   1. Myocardial infarction or stroke/transient ischemic attack within the 6 months prior to study entry.
   2. Uncontrolled angina within the 3 months prior to study entry.
   3. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes, or poorly controlled atrial fibrillation).
   4. Corrected QT (QTc) prolongation > 480 msec.
   5. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled venous thrombus).
   6. Cardiovascular disease-related requirement for daily supplemental oxygen.
   7. History of two or more myocardial infarction or two or more coronary revascularization procedures.
   8. Subjects with history of myocarditis, regardless of etiology.
   9. Troponin T (TnT) or I (TnI) > ULN.
10. Subjects with history of life-threatening toxicity related to prior immune therapy (eg. anti-cytotoxic T-lymphocyte-associated protein [CTLA]-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg, hormone replacement after endocrinopathy).
11. Active or prior documented inflammatory bowel disease (e.g. crohn disease, ulcerative colitis),
12. Current or prior use of immunosuppressive medication within 28 days before the first dose of nivolumab, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent (use for brain metastases is not permitted 28 days prior to start of therapy).
13. Active or prior documented autoimmune disease within the past 3 years. Note: Subjects with active, known or suspected autoimmune disease such as vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
14. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment,
15. History of idiopathic pulmonary fibrosis, history of non-infectious pneumonitis that required steroids, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted,
16. Has an active neurological disease, as well as an history of encephalitis, meningitis or uncontrolled seizures in the 12 months prior to study entry,
17. Has en history of myocarditis,
18. Has known active hepatitis B or hepatitis C,
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV1/2 antibodies),
20. Has a known history of tuberculosis,
21. Participant with oral anticoagulation therapy,
22. Prior organ transplantation, including allogeneic stem cell transplantation,
23. Has an active infection requiring systemic treatment within two weeks prior study entry,
24. Has received a live vaccine within 30 days prior to the first dose of trial treatment,
25. Individuals deprived of liberty or placed under legual guardianship,
26. Body weight < 40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of nivolumab in association with relatlimab independently for each arm | 6 months
  Antitumor activity will be assessed in terms of 6-month progression-free rate and is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), based on RECIST 1.1

SECONDARY OUTCOMES:
Best overall response, independently for each arm | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determined once all the data for the patient is known (RECIST 1.1)
1-year progression-free survival, independently for each arm | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
2-year progression-free survival, independently for each arm | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
1-year overall survival, independently for each arm | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause)
2-year overall survival, independently for each arm | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause)
Growth Modulation Index, independently for each arm | throughout the treatment period, an expected average of 6 months
  GMI is defined for each patient as the ratio of its PFS on the nivolumab + relatlimab treatment combination to its PFS on the previous line of therapy (Von Hoff 1998)
Safety profile, independently for each arm | throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Blood cytokines levels | baseline, cycle 1 day 1, cycle 1 day 15, cycle 3 day 1 and progression (each cycle is 28 days)
  Levels of cytokines in blood will be measured by ELISA
Blood lymphocytes levels | baseline, cycle 1 day 1, cycle 1 day 15, cycle 3 day 1 and progression (each cycle is 28 days)
  Levels of lymphocytes in blood will be measured by flow cytometry
Blood kynurenine levels | baseline, cycle 1 day 1, cycle 1 day 15, cycle 3 day 1 and progression (each cycle is 28 days)
  Levels of kynurenine in blood will be measured by ELISA
Tumor immune cells levels | before treatment onset and cycle 3 day 1 (each cycle is 28 days)
  Levels of immune cells in tumor will be measured by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Nantes
  - Hôpital Cochin, Paris
  - Institut Gustave Roussy, Villejuif